CLINICAL TRIAL: NCT02846077
Title: Multi-scale Modeling of Sleep Behaviors in Social Networks
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Elizabeth B. Klerman, Associate Professor, Brigham and Women's Hospital
Other Study IDs: BrighamHospital
Record Dates: First submitted 2016-07-15; First posted 2016-07-27 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Healthy Volunteers
Keywords: sleep; social networks; undergraduates; mood; circadian rhythms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- College students: College students will be monitored and will complete online surveys, install apps on their mobile phones, wear physiological sensors and provide saliva samples for later assay.
  Interventions: Other: No intervention. Observation only

INTERVENTIONS:
Other: No intervention. Observation only — No intervention. Observation only

SUMMARY:
The project is designed to document in college undergraduates the relationships among sleep/wake timing and duration, use of mobile phones and other electronic devices, food timing and content, self-reported mood and physiological measures.

DETAILED DESCRIPTION:
College undergraduates are studied in cohorts of ~ 50 in fall or spring semesters. They complete diaries once in the morning and once in the evening about sleep/wake timing, timing of social and school activities, and mood. They wear physiological sensors. They install (1) an application on their mobile phone that tracks timing, duration and de-identified sender/recipient of phone calls and text messages, use of internet or apps (but not the content or names of those internet sites and apps) and (2) meal content and timing. They also spend at least one overnight session providing saliva samples for later assay for hormones.

ELIGIBILITY:
Inclusion Criteria:

* undergraduate at institution at which we have permission to perform study
* owning a mobile device on which the phone app can be installed
* ability to wear the wrist-worn sensors

Exclusion Criteria:

* no travel outside one time zone starting approximately 2 weeks before monitoring begins through end of approximately one month of monitoring.
* participation in a prior group studied

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: College undergraduates
Sampling Method: Non-Probability Sample
Enrollment: 729 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Timing of sleep and wake | Approximately one month
  Timing of self-reported sleep onset and wake onset
Timing of phone use (e.g., mobile phone calls, text messages, applications and internet use) | Approximately one month
  Timing of phone use (e.g, mobile phone calls, text messages, applications and internet use)

SECONDARY OUTCOMES:
Mood | Approximately one month
  Self-reported mood using a linear non-numeric scale
Activity levels | approximately one month
  Activity levels collected every minute using a wrist-worn device
Light exposure levels | approximately one month
  Light exposure levels collected every minute using a wrist-worn device
Food choice | approximately one month
  Content of food
Circadian phase | one day
  Calculated time of melatonin phase as a marker of circadian rhythms
Electrodermal activity | approximately one month
  Electrodermal activity as measured using a wrist-worn device
Timing of meals | approximately one month
  Time meals are eaten

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Klerman, MD PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lu S, Stone JE, Klerman EB, McHill AW, Barger LK, Robbins R, Fischer D, Sano A, Czeisler CA, Rajaratnam SMW, Phillips AJK. The organization of sleep-wake patterns around daily schedules in college students. Sleep. 2024 Sep 9;47(9):zsad278. doi: 10.1093/sleep/zsad278. PMID 37930792
- [Derived] Khalid M, Sano A. Exploiting social graph networks for emotion prediction. Sci Rep. 2023 Apr 13;13(1):6069. doi: 10.1038/s41598-023-32825-9. PMID 37055459
- [Derived] Fischer D, McHill AW, Sano A, Picard RW, Barger LK, Czeisler CA, Klerman EB, Phillips AJK. Irregular sleep and event schedules are associated with poorer self-reported well-being in US college students. Sleep. 2020 Jun 15;43(6):zsz300. doi: 10.1093/sleep/zsz300. PMID 31837266
- [Derived] McHill AW, Phillips AJ, Czeisler CA, Keating L, Yee K, Barger LK, Garaulet M, Scheer FA, Klerman EB. Later circadian timing of food intake is associated with increased body fat. Am J Clin Nutr. 2017 Nov;106(5):1213-1219. doi: 10.3945/ajcn.117.161588. Epub 2017 Sep 6. PMID 28877894